CLINICAL TRIAL: NCT06549868
Title: Using Yoga to Reduce Chaos and Improve Preschooler Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Guseman (Other)
Responsible Party: Sponsor-Investigator, Emily Guseman, Assistant Professor, Ohio University College of Osteopathic Medicine
Organization: Ohio University College of Osteopathic Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-X-124
Record Dates: First submitted 2024-07-24; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Sleep, Inadequate; Sleep
Keywords: sleep; children; preschool; yoga; parents; household chaos
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Participants will be asked to follow a yoga-based bedtime routine for 4 weeks
  Interventions: Behavioral: Yoga-based bedtime routine
- Story (Other): Waitlist control arm. Participants will complete a 4-week control period upon randomization. After this control period is completed, they will crossover into the intervention group and follow the same 4 week intervention as the yoga group.
  Interventions: Behavioral: Yoga-based bedtime routine

INTERVENTIONS:
Behavioral: Yoga-based bedtime routine — Dyads in the yoga intervention group receive a picture book outlining a bedtime-themed yoga routine and are instructed to incorporate it into their bedtime routine at least four nights per week for four weeks. The routine guides children through a sequence of yoga poses, starting with the mountain pose and ending in child's pose, designed to calm them as the story progresses. Parents are given a bedtime diary to record the date, whether the child completed the yoga routine each evening, and any comments about their experience with the book.
  At week 6, families return to the lab, complete anthropometric assessments and questionnaires, and are fitted with accelerometers to wear for the next week. The accelerometers are returned and data is downloaded a week later. Families are then encouraged to continue using the yoga routine as often as they wish for an additional four weeks, although the frequency of use is not tracked during this maintenance period.

SUMMARY:
The goal of this intervention study is to learn if a yoga-based bedtime routine is feasible for families to follow and to learn if the routine is effective at improving preschooler sleep. The main question it aims to answer is:

Will families be able to follow the routine regularly during the study period? Will following the yoga routine improve household chaos and preschooler sleep? Researchers will compare the yoga group to a control group to see if implementing the yoga routine works better than simple advice to read a bedtime story.

Participants will be asked to visit the lab 4 times. At the first visit, we will measure body size of parents and children, ask parents to complete some surveys, and fit each of them with an activity monitor. One week later, they will return for the second visit. At this visit, we will collect the activity monitor and assign the participants to either the intervention (yoga) or control (bedtime story) group. Families in the intervention group will learn about the intervention and be asked to follow it for the next four weeks. Families in the control group will receive a book and advice about reading stories at bedtime. After four weeks, families will return to the lab for a third visit and we will repeat the measurements from visit 1. Then, families in the intervention group will be asked to follow the yoga routine as much as they would like to for the next 4 weeks. Families in the control group will "cross over" to the intervention group and will follow the yoga intervention for 4 weeks. Then, families will return to the lab for a 4th visit, where we will repeat all of the measures from the first visit and the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2.0-5.9 years of age and their self-identified primary parent/guardian

Exclusion Criteria:

- Parent currently pregnant Child or parent unable to walk independently Child or parent has an upper body mobility limitation that precludes completion of yoga routine

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Intervention adherence | 4 weeks
  Number of yoga sessions completed Percent of prescribed sessions completed
Household chaos | at week 1, week 5, and week 10
  Measured using Chaos, Hubbub, and Order Scale (CHAOS) at enrollment, crossover point, and study completion. A lower CHAOS score post-intervention would indicate an improvement in household chaos.

SECONDARY OUTCOMES:
Child sleep duration | at week 1, week 5, and week 10
  nightly sleep measured by waist-worn accelerometer at enrollment, crossover point, and study completion
Parent sleep duration | 1 week at week 1, week 5, and week 10
  nightly sleep measured by waist-worn accelerometer at enrollment, crossover point, and study completion
Parent sleep quality | 1 week at week 1, week 5, and week 10
  nightly sleep measured by waist-worn accelerometer at enrollment, crossover point, and study completion
Child sleep quality | 1 week at week 1, week 5, and week 10
  nightly sleep measured by waist-worn accelerometer
Child sleep quality | 1 week at week 1, week 5, and week 10
  measured by Children's Sleep Habits Questionnaire (CSHQ; scored using mean and standard deviation of survey items. A higher CSHQ mean score indicates worse sleep quality)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study for a planned full-scale intervention